CLINICAL TRIAL: NCT00278070
Title: Metronomic Vinorelbine in Patients With Metastatic Tumors: Phase II Translational Study
Brief Title: Metronomic Oral Vinorelbine in Patients With Metastatic Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Cooperative Oncology Group (Other)
Collaborators: University of Ioannina (Other)
Responsible Party: Evangelos Briasoulis, Hellenic Cooperative Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE 50/05
Record Dates: First submitted 2006-01-17; First posted 2006-01-18 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Breast Cancer; Non Small Cell Lung Cancer; Prostate Cancer
Keywords: Metronomic-therapy; vinorelbine; Recurrent Breast Cancer; Recurrent Non Small Cell Lung Cancer; Metastatic prostate cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: vinorelbine oral formulation
- 2 (Active Comparator)
  Interventions: Drug: vinorelbine oral formulation
- 3 (Active Comparator)
  Interventions: Drug: vinorelbine oral formulation

INTERVENTIONS:
Drug: vinorelbine oral formulation — Patients will take three times a week [Monday, Wednesday and Friday] by mouth, a standard dose of soft capsules of vinorelbine given at dose ascribed by randomization procedure
  Other Names: Navelbine

SUMMARY:
Patients with recurrent or metastatic solid tumors receive oral vinorelbine at one of three different doses (30 or 40 or 50 mg). Vinorelbine will be administered orally at a metronomic schedule three times a week: on Monday, Wednesday and Friday.

DETAILED DESCRIPTION:
The purpose of this study is to define the biologically optimal dose of vinorelbine when administered at a metronomic dosing schema. [Metronomic chemotherapy refers to the close, regular administration of minimally toxic doses of cytotoxic drugs, with minimal or no drug-free breaks, over prolonged periods]. Patients with recurrent or metastatic solid tumors are randomly assigned one of three different doses of oral vinorelbine (30 or 40 or 50 mg). Treatment is administered three times a week (Monday, Wednesday and Friday) continuously until disease progression or unacceptable toxicity or to a maximum of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Ages 16 - 75 years
* Genders: both
* Performance status 0-2 according to the World Health Organization (WHO) scale
* Life expectancy of at least 16 weeks
* Adequate bone marrow, hepatic and renal functions
* Absence of brain metastasis
* Metastatic/locally advanced refractory prostate, breast or non-small cell lung cancer previously treated with no more than two chemotherapeutic regimens
* White blood cells >= 3500/mm^3
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Total serum bilirubin less than 1.5 mg/dl
* Serum transaminases less than 2.0 x upper normal limit (UNL) unless attributed to liver metastases
* Serum creatinine within normal range

Exclusion Criteria:

* Major active infection
* More than two prior chemotherapy regimens for metastatic disease
* Any of the following within the 12 months prior to starting the study treatment:

  * myocardial infarction,
  * severe/unstable angina,
  * coronary/peripheral artery bypass graft,
  * congestive heart failure,
  * cerebrovascular accident or transient ischemic attack, or pulmonary embolism,
  * cardiac dysrhythmias of grade >/= 2,
  * atrial fibrillation of any grade, or
  * heart rate corrected interval (QTc) > 450 msec for males or > 470 msec for females.
* Hypertension that cannot be controlled with medications (> 150/100 mmHg despite optimal medical therapy)
* Ongoing anti-coagulation therapy
* Pregnancy or breastfeeding
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration; or which, in the judgment of the investigator, would make the patient inappropriate for entry into the trial.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-01; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
time to treatment failure | TTF rates per arm will be compared at 4 and 6 months

SECONDARY OUTCOMES:
progression free survival | Patients will be assessed every 2 months during the first 6 months on treatment and every 4 months thereafter until documentation of objective tumor progression or death.
time to progression | Patients will be assessed every 2 months during the first 6 months on treatment and every 4 months thereafter until documentation of objective tumor progression.
toxicity | Acute toxicity will be assessed during the first 8 weeks, sub-acute 8 weeks to 4 months, chronic post 4 months
changes in blood concentrations of angiogenesis-associated surrogate markers and pharmacokinetics | Baseline values will be assessed for predictive potential and assessment on weeks 2,4,8, 12 and thereafter every 2 months they will be analyzed for their capacity to act as surrogate markers of treatment activity

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Briasoulis, MD, Principal Investigator — Assistant Professor of Oncology, Medical School, University of Ioannina
Locations (11):
- Greece (11):
  - Henry Dunant Hospital, Athens
  - Sotiria Hospital, Athens
  - University Hospital "Attikon", Athens
  - Agii Anargiri Cancer Hospital, Athens
  - Hygeia Hospital, Athens
  - Metropolitan Hospital, Athens
  - General Hospital of Chania, Chania
  - University General Hospital of Ioannina, Medical Oncology Dept, Ioannina
  - University Hospital of Patras, Pátrai
  - "Theagenio" Hospital, Thessaloniki
  - "Papageorgiou" Cancer Hospital, Thessaloniki

REFERENCES:
- [Derived] Briasoulis E, Aravantinos G, Kouvatseas G, Pappas P, Biziota E, Sainis I, Makatsoris T, Varthalitis I, Xanthakis I, Vassias A, Klouvas G, Boukovinas I, Fountzilas G, Syrigos KN, Kalofonos H, Samantas E. Dose selection trial of metronomic oral vinorelbine monotherapy in patients with metastatic cancer: a hellenic cooperative oncology group clinical translational study. BMC Cancer. 2013 May 29;13:263. doi: 10.1186/1471-2407-13-263. PMID 23718900